CLINICAL TRIAL: NCT03980951
Title: A Randomized Comparison of Epidural, Dural Puncture Epidural and Combined Spinal Epidural Without Intrathecal Opioids for Labor Analgesia.
Brief Title: Neuroaxial Labour Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: elite medical hospital (Unknown)
Responsible Party: Sponsor-Investigator, Wahba bakhet, Director, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019 WB
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Labor Analgesia
MeSH Terms: interventions — Injections, Epidural

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial assignment placed in sealed envelopes.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- combined spinal epidural group (Active Comparator): Bupivacaine 2.5 mg
  Interventions: Procedure: Combined Spinal Epidural without intrathecal opioids
- dura puncture epidural group (Active Comparator): Bupivacaine 0.125% with Fentanyl 2 mcg/mL, 20 mL load over 5 min
  Interventions: Procedure: Dural Puncture Epidural Technique
- epidural (Active Comparator): Bupivacaine 0.125% with Fentanyl 2 mcg/mL, 20 mL load over 5 min
  Interventions: Procedure: epidural

INTERVENTIONS:
Procedure: Dural Puncture Epidural Technique — three labor analgesia techniques
  Arms: dura puncture epidural group
Procedure: Combined Spinal Epidural without intrathecal opioids — three labor analgesia techniques
  Arms: combined spinal epidural group
Procedure: epidural — three labor analgesia techniques
  Arms: epidural

SUMMARY:
The primary outcome of this clinical trial is to compare the pain scores during labour and delivery of combined spinal epidural without intrathecal opioids and dural puncture epidural

The secondary objective of this study is to compare the and fetomaternal outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous parturient
2. Singleton, vertex gestation at term (37-42 weeks)
3. Less than 5 cm dilation
4. request an epidural technique for labor analgesia

Exclusion Criteria:

1. Hypersensitivity to local the study drugs
2. Clinically significant disease , including diseases of pregnancy (i.e preeclampsia, gestational diabetes)
3. Any contraindication to the administration of an epidural technique
4. Risk factor for cesarean delivery.
5. fetal anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females requesting labor analgesia
Enrollment: 120 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
epidural Local anesthetic consumption | 1 year

SECONDARY OUTCOMES:
Maternal hypotension | 1 year
  maternal mean arterial blood pressure less than 50 mmhg
incidence of fetal bradycardia | 1 year
  a fetal heart rate of less than 100 beats per minute
incidence of maternal pruritus | 1 year
  Participants will be assessed for pruritus every hour, by grading the severity on a scale ranging from 0-3; 0 = none, 1 = mild, 2= moderate and 3 = severe
labour pain scores | 1 year
  Visual analogue scale with its 0 to 10 score range: (0 (no pain) to 10 ( Severe pain)

CONTACTS AND LOCATIONS:
Locations (2):
- Ain Shams University, Cairo, Abbasyia, Egypt
- Elite Hospital, Kuwait City, Abbasyia, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakhet WZ. A randomized comparison of epidural, dural puncture epidural, and combined spinal-epidural without intrathecal opioids for labor analgesia. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):231-236. doi: 10.4103/joacp.JOACP_347_19. Epub 2021 Jul 15. PMID 34349372